CLINICAL TRIAL: NCT00705510
Title: Efficacy of 0.05 % Cyclosporine Ophthalmic Emulsion Compare With Tear in Meibomian Gland Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Pinnita Prabhasawat, Department of Ophthalmology; Siriraj Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 154/2551(EC1)
Record Dates: First submitted 2008-06-24; First posted 2008-06-26 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2010-11

CONDITIONS: Meibomian Gland Dysfunction
Keywords: Cyclosporine; Unstable tear film; Meibomian gland; Meibomian gland dysfunction
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: 0.05% cyclosporin eye drop
- B (Placebo Comparator)
  Interventions: Drug: 0.05% cyclosporin eye drop

INTERVENTIONS:
Drug: 0.05% cyclosporin eye drop — use the medication twice daily for 3 months
  Other Names: Restasis eye drop, Cellufresh eye drop

SUMMARY:
To evaluate the efficacy of 0.05% cyclosporine ophthalmic emulsion (Restasis® , Allergan) versus an artificial tears alone in patients with meibomian gland dysfunction that have abnormal tear quality and quantity by subjective symptoms and signs including tear breakup time

DETAILED DESCRIPTION:
Meibomian gland dysfunction patients will divide into 2 groups. One group will have 0.05% cyclosporine opthalmic emulsion and the other will have non-preservative artificial tear twice daily, compare the result in 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, of legal age of consent
* Patient has a diagnosis of meibomian gland dysfunction with at least 1 symptom as the following; ocular burning, ocular discomfort, and grittiness
* Had a slit-lamp diagnosis of meibomian gland dysfunction based on the presence of one of the following

  * meibomian gland inflammation by lid margin or tarsal erythema, bulbar conjunctiva hyperemia, telangiectasia or thickening irregularity of the eyelid margins
  * meibomian gland orifice inclusion (plugging) or abnormal of secretion
* Non-invasive tear break up time (NTBUT) with Tear scope Plus(Keeler, Windsor, UK) ≤ 8 seconds
* Ability to follow study instruction and likely to complete all required visits

Exclusion Criteria:

* Age < 18 years old
* Patients with severe ocular disease from Steven Johnson syndrome burn, limbal deficiency
* Patients used cyclosporine within past 1 year
* Patients used oral cyclosporine or anticholinergic drug within past 2 months
* Patients with HIV or autoimmune disease
* Patients with active ocular infections and patients with a history of herpes keratitis
* Patients with known or suspected hypersensitivity to any of the ingredients in the formula (cyclosporine, glycerin, castor oil, polysorbate 80, carbomer 1342)
* Female patients are pregnant or nursing
* Patients who wear contact lenses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
NTBUT | 0,1,2,3 month

SECONDARY OUTCOMES:
OSDI score, FTBUT, lid inflammation, meibomian gland secretion and expressibility, bulbar and tarsal conjunctival injection,fluorescein staining, rose bengal staining | 0,1,2,3 month

CONTACTS AND LOCATIONS:
Overall Officials: Pinnita Prabhasawat, MD, Principal Investigator — Department of Ophthalmology, Siriraj H, Mahidol U
Locations (1):
- Department of Ophthalmology; Siriraj Hospital, Bangkok, Bangkok, Thailand